CLINICAL TRIAL: NCT00637923
Title: Phase II, Randomized, Double-blind, Placebo-controlled Study of Nitazoxanide in Combination With Peginterferon Alfa-2a and Ribavirin in Treatment-Naive Patients With Hepatitis C
Brief Title: Study of Nitazoxanide, Peginterferon Alfa-2a and Ribavirin in Treatment-Naive Hepatitis C Patients
Acronym: STEALTHC-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM01-2026
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — nitazoxanide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): One nitazoxanide 500 mg tablet orally with food twice daily (b.i.d.) for 4 weeks followed by 500 mg nitazoxanide b.i.d. plus one weekly injection of 180µg of peginterferon α-2a plus weight-based ribavirin for 48 weeks.
  Interventions: Drug: Nitazoxanide; Biological: Peginterferon alfa-2a; Drug: Ribavirin
- 2 (Placebo Comparator): One placebo tablet orally with food twice daily (b.i.d.) for 4 weeks followed by placebo b.i.d. plus one weekly injection of 180µg of peginterferon α-2a plus weight-based ribavirin for 48 weeks.
  Interventions: Drug: Placebo; Biological: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Nitazoxanide — One nitazoxanide 500 mg tablet orally with food twice daily (b.i.d.) for 4 weeks followed by 500 mg nitazoxanide b.i.d. plus one weekly injection of 180µg of peginterferon α-2a plus weight-based ribavirin for 48 weeks.
  Other Names: Alinia
  Arms: 1
Drug: Placebo — One placebo tablet orally with food twice daily (b.i.d.) for 4 weeks followed by placebo b.i.d. plus one weekly injection of 180µg of peginterferon α-2a plus weight-based ribavirin for 48 weeks.
  Arms: 2
Biological: Peginterferon alfa-2a — One weekly injection of 180µg of peginterferon α-2a for 48 weeks.
  Other Names: PEGASYS
Drug: Ribavirin — Weight-based ribavirin for 48 weeks.
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to determine if nitazoxanide in combination with peginterferon alfa-2a and ribavirin is safe and effective in treating chronic hepatitis C in treatment-naive patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C genotype 1.

Exclusion Criteria:

* Patients that have previously received treatment with any interferon or interferon-based treatment for chronic hepatitis C.
* Females of child-bearing age who are either pregnant, breast-feeding or not using birth control and are sexually active.
* Males whose female partners are either pregnant or of child-bearing potential or not using birth control and are sexually active.
* Other causes of liver disease including autoimmune hepatitis.
* Transplant recipients receiving immune suppression therapy.
* Screening tests positive for Anti-Hepatitis A Virus Immunoglobulin M Antibody (anti-HAV IgM Ab), Hepatitis B's antigen (HBsAg), Anti-Hepatitis B core Immunoglobulin M Antibody (anti-HBc IgM Ab) or Anti-Human Immunodeficiency Virus Antibody (anti-HIV Ab).
* Decompensated cirrhosis, history of variceal bleeding, ascites, hepatic encephalopathy, Child-Turcotte-Pugh (CTP) score >6 or Model for End-stage Liver Disease (MELD) score >8.
* Alcohol consumption of >40 grams per day or an alcohol use pattern that will interfere with the study.
* Absolute neutrophil count <1500 cells/mm3; platelet count <135,000 cells/mm3; hemoglobin <12 g/dL for women and <13 g/dL for men; or serum creatinine concentration ≥1.5 times Upper Limit of Normal (ULN).
* Hypothyroidism or hyperthyroidism not effectively treated with medication.
* Hemoglobin A1C (HgbA1c) >7.5 or history of diabetes mellitus.
* Body Mass Index (BMI) >34.
* History or other clinical evidence of significant or unstable cardiac disease.
* History or other clinical evidence of chronic pulmonary disease associated with functional impairment.
* Serious or severe bacterial infection(s).
* Ulcerative or hemorrhagic/ischemic colitis.
* Pancreatitis.
* History of severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization.
* History of uncontrolled severe seizure disorder.
* Requires concomitant theophylline or methadone.
* History of immunologically mediated disease requiring more than intermittent anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids.
* History or other evidence of severe retinopathy or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension.
* Hemoglobinopathies.
* History of hypersensitivity or intolerance to nitazoxanide or any of the excipients comprising the nitazoxanide tablets, peginterferon alfa-2a injectable solution or ribavirin tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmet B Keeffe, MD, MACP, Study Director — Romark Laboratories L.C.; Norman Gitlin, MD, Principal Investigator — Atlanta Gastroenterology Associates; Joseph K Lim, MD, Principal Investigator — Yale University; Ira Jacobson, MD, Principal Investigator — New York Presbyterial-Weill Medical College of Cornell University; Mitchell L Shiffman, MD, Principal Investigator — McGuire Veteran's Administration Medical Center; Ronald E Pruitt, MD, Principal Investigator — Nashville Medical Research Institute; Arthur Berman, DO, Principal Investigator — Florida Center for Gastroenterology; Bruce Bacon, MD, Principal Investigator — St. Louis University Medical Center; Nezam Afdhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center; David Johnson, MD, Principal Investigator — Bay Pines VA Healthcare System; Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital; Vinod Rustgi, MD, Principal Investigator — Metropolitan Research; Aijaz Ahmed, MD, Principal Investigator — Stanford University
Locations (10):
- United States (10):
  - Palo Alto VA Healthcare System, Palo Alto, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York Presbyterian-Weill Medical College of Cornell University, New York, New York
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Metropolitan Research, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients from 13 study centers in the United States, including 2 Veterans Administration hospitals.
Groups:
- NTZ+PR: One nitazoxanide 500 mg tablet orally with food twice daily (b.i.d.) for 4 weeks followed by 500 mg nitazoxanide b.i.d. plus one weekly injection of 180µg of peginterferon α-2a plus weight-based ribavirin for 48 weeks.
- Placebo+PR: One placebo tablet orally with food twice daily (b.i.d.) for 4 weeks followed by placebo b.i.d. plus one weekly injection of 180µg of peginterferon α-2a plus weight-based ribavirin for 48 weeks.
Period: Overall Study
Arm/Group | NTZ+PR | Placebo+PR
Started | 75 | 37
Completed | 45 | 18
Not Completed | 30 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NTZ+PR | Placebo+PR | Total
Number analyzed (Participants) | 75 | 37 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 37 | 111
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7) | 51 (8) | 50 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 13 | 39
  Male | 49 | 24 | 73
Region of Enrollment [Number; unit: participants]
  United States | 75 | 37 | 112

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection 24 weeks after the end of treatment. All others were considered non-responders.
Time Frame: 24 weeks after end of treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 75 | 37
participants
  Responders | 32 | 13
  Non-responders | 43 | 24

2. Secondary Outcome: End of Treatment Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection at the end of treatment. All others were considered non-responders.
Time Frame: At end of treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 75 | 37
participants
  Responders | 46 | 18
  Non-responders | 29 | 19

3. Secondary Outcome: Early Virologic Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection after 12 weeks of combination therapy.
Time Frame: After 12 weeks combination treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 75 | 37
participants
  Responders | 45 | 18
  Non-responders | 30 | 19

4. Secondary Outcome: Rapid Virologic Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection after 4 weeks of combination therapy.
Time Frame: After 4 weeks combination treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 75 | 37
participants
  Responders | 9 | 7
  Non-responders | 66 | 30

5. Secondary Outcome: Changes in ALT
Description: This analysis was conducted using a comparison of changes in Alanine aminotransferase (ALT) from baseline through week 8, week 16, end of treatment and end of follow up.
Time Frame: From baseline to week 8
Population: This analysis was conducted using only data for patients that completed the baseline through week 8 time points.
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 71 | 35
participants
  Remains Elevated | 23 | 5
  Elevated to Normal | 29 | 11
  Remains Normal | 16 | 17
  Normal to Elevated | 3 | 2

6. Secondary Outcome: Changes in ALT
Description: as for outcome 5
Time Frame: From baseline to week 16
Population: This analysis was conducted using only data for patients that completed the baseline through week 16 time points.
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 68 | 31
participants
  Remains Elevated | 12 | 4
  Elevated to Normal | 38 | 11
  Remains Normal | 17 | 15
  Normal to Elevated | 1 | 1

7. Secondary Outcome: Changes in ALT
Description: as for outcome 5
Time Frame: From baseline to end of treatment
Population: This analysis was conducted using only data for patients that completed the baseline through end of treatment time points.
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 45 | 18
participants
  Remains Elevated | 4 | 3
  Elevated to Normal | 28 | 6
  Remains Normal | 13 | 9
  Normal to Elevated | 0 | 0

8. Secondary Outcome: Changes in ALT
Description: as for outcome 5
Time Frame: From baseline to end of follow up
Population: This analysis was conducted using only data for patients that completed the baseline through the end of follow-up time points.
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 45 | 18
participants
  Remains Elevated | 9 | 2
  Elevated to Normal | 23 | 7
  Remains Normal | 13 | 8
  Normal to Elevated | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Arm/Group | NTZ+PR | Placebo+PR
Serious Adverse Events (participants affected / at risk) | 12/75 | 7/37
Other Adverse Events (participants affected / at risk) | 73/75 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTZ+PR (N=75) | Placebo+PR (N=37)
PAIN ABDO (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
RETINAL DIS (Eye disorders) | 1 (1) | 0 (0)
CARCINOMA LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
GASTROENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PNEUMONIA ASPIR (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INFARCT MYOCARD (Cardiac disorders) | 1 (1) | 0 (0)
KIDNEY FAIL (Renal and urinary disorders) | 1 (1) | 1 (1)
DEHYDRAT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CONSTIP (Gastrointestinal disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
BONE FRACT SPONTAN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HYPOKALEM (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HEM GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
HYPERTENS (Vascular disorders) | 0 (0) | 1 (1)
FEVER (General disorders) | 0 (0) | 1 (1)
EFFUS PLEURAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
APNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HEART ARREST (Cardiac disorders) | 0 (0) | 1 (1)
EMOTION LABIL (Nervous system disorders) | 0 (0) | 1 (1)
HYPERKALEM (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTZ+PR (N=75) | Placebo+PR (N=37)
Diarrhea (Gastrointestinal disorders) | 36 (36) | 8 (8)
Nausea (Gastrointestinal disorders) | 32 (32) | 10 (10)
Anorexia (Gastrointestinal disorders) | 21 (21) | 4 (4)
Stomatitis Ulcer (Gastrointestinal disorders) | 10 (10) | 2 (2)
Vomit (Gastrointestinal disorders) | 9 (9) | 1 (1)
Constip (Gastrointestinal disorders) | 9 (9) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 6 (6)
Asthenia (General disorders) | 52 (52) | 25 (25)
Headache (General disorders) | 26 (26) | 15 (15)
Pain (General disorders) | 22 (22) | 7 (7)
Fever (General disorders) | 15 (15) | 6 (6)
Pain Abdo (Gastrointestinal disorders) | 12 (12) | 6 (6)
Chills (General disorders) | 11 (11) | 4 (4)
Inject site react (General disorders) | 9 (9) | 2 (2)
Flu Synd (General disorders) | 6 (6) | 4 (4)
Insomnia (Nervous system disorders) | 27 (27) | 10 (10)
Nervousness (Nervous system disorders) | 24 (24) | 6 (6)
Depression (Nervous system disorders) | 22 (22) | 9 (9)
Thinking Abnorm (Nervous system disorders) | 16 (16) | 6 (6)
Dizziness (Nervous system disorders) | 12 (12) | 6 (6)
Emotion labil (Nervous system disorders) | 10 (10) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 37 (37) | 11 (11)
Pruritis (Skin and subcutaneous tissue disorders) | 24 (24) | 8 (8)
Skin dry (Skin and subcutaneous tissue disorders) | 21 (21) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (19) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 12 (12)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 8 (8)
Cough inc (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 4 (4)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Urin Abnorm (Renal and urinary disorders) | 32 (32) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 30 (30) | 11 (11)
Leukopenia (Blood and lymphatic system disorders) | 16 (16) | 10 (10)
Weight dec (Metabolism and nutrition disorders) | 12 (12) | 6 (6)
Hypercholesterem (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 9 (9)
Hypertens (Vascular disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Presentation and/or publication is encouraged provided the Sponsor is notified in advance and given the opportunity to review the manuscript or abstract 30 days prior to its submission for presentation at a scientific meeting or for publication in a scientific journal. The investigators will have complete autonomy regarding the content and wording including the decision of whether or not to publish.